CLINICAL TRIAL: NCT02928172
Title: Monitoring the Responses to Nociceptive Stimuli During General Anesthesia Based on Electroencephalographic Signals, an Observational Study
Brief Title: Comparison of Two Electroencephalograms (EEG) Monitors in Patients Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00043738
Record Dates: First submitted 2016-10-04; First posted 2016-10-10 (Estimated); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Deep Sedation
Keywords: q-CON; q-NOX; BIS; Electroencephalograms (EEG); Laryngeal Mask Airway (LMA); Sedation; General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Depth of Anesthesia (Other): Subjects will have the qCON-qNOX and BIS monitor
  Interventions: Device: qCON-qNOX; Device: BIS

INTERVENTIONS:
Device: qCON-qNOX — Each subject will have the qCON-qNOX monitor on his/her forehead + the BIS monitor
Device: BIS — Each subject will have the BIS monitor on his/her forehead + the qCON-qNOX monitor

SUMMARY:
Hypothesis:

There is a statistically measurable correlation between qNOX and rough clinical signs of insufficient anti-nociception such as movements during Laryngeal Mask Airway (LMA) insertion, skin Incision, LMA removal. It will reduce the problem of anticipating the nociception in patients undergoing general anesthesia.

Objectives:

1. to compare two indexes of hypnosis, the qCON (Quantium Medical, Spain) with the Bispectral index (BIS™) (Covidien, Boulder CO. USA), in patients undergoing surgery under sedation and general anesthesia.
2. to assess the qNOX index of pain/nociception (Quantium Medical, Barcelona, Spain) and the qCON index of hypnosis.
3. to assess qNOX reliability as a specific indicator of response to nociceptive stimulation.

DETAILED DESCRIPTION:
Monitoring the anti-nociceptive drug effect is useful because a sudden and strong nociceptive stimulus may result in untoward autonomic responses and muscular reflex movements. Unopposed stimulation may also 'overrule' a state of stable unconsciousness, with resultant awakening and awareness. The traditional clinical use of systolic or mean blood pressure is actually still one of the methods in everyday use for this monitoring purpose. Another cornerstone is the experience of which drugs and doses are effective in attenuating nociception. Alpiger and colleagues found that simple end-tidal monitoring of sevoflurane was a better predictor of nociceptive response than Auditory Evoked Potential.

Thus, monitoring the state of anti-nociception with objective, non-clinical methods is still in a state of testing and development, without well-documented and proven methods for consistent 'no-fuss' clinical daily use. Some methods, like those using systolic blood pressure, are based on the reduced sympathetic response from the Central Nervous System (CNS) when in a state of drug-induced anti-nociception during concomitant surgical stress. These include the pulse plethysmogram amplitude, heart rate variability and/or amplitude, pupillometry, muscle tonus and skin conductance.They all have limitations in interpretation, as the state of sympathetic tone is strongly influenced by numerous factors, including hypovolemia, vasopressors, atropine and patient positioning. In addition, sympathetic tone is very unspecific in the awake or lightly sedated patient, as mood and subjective feelings have a strong impact.

Attempts are also been made on using the EEG for monitoring of anti-nociception. This approach has been challenged as difficult, as most of the antinociceptive drugs effects are in the periphery, the medullary cord or deeper cerebral layers, far from the EEG signals derived from the frontal cortex. However, EEG is a 'mirror' of what is going on in other parts of the CNS and peripheral nervous system. One problem is to elucidate how the EEG signals may be used in a sensitive and specific way to reflect anti-nociception. Concepts such as response-entropy, Composite Variability Index and BIS variability score have been tested and launched.

Quantium Medical has an EEG-based algorithm with two outputs: the qCON for unconsciousness and the qNOX for anti-nociception. This means that calculates and displays two indices. One, the qCON, is designed to provide information about the depth of the hypnotic state, similar to that provided by the BIS™ and Sedline™ monitor (Masimo, Irvine CA). The second index, the qNOX, is designed to provide information about the depth of the antinociceptive state. The qCON has shown a comparable performance with BIS, and qNOX has proved correlation with rough clinical signs of insufficient antinociception, such as movements during LMA insertion, laryngoscopy and tracheal intubation

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo general surgical procedures with general anesthesia/LMA.
* Willingness and ability to sign an informed consent document.
* 18 - 80 years of age.
* ASA Class I - III adults of either sex

Exclusion Criteria:

* Inability to consent
* Withdrawal criteria
* Electrodes should be changed when patient's skin impedance value exceeds 15 kΩ after conditioning skin properly. If after two changes of electrodes, impedance remains above 15 kΩ, patient will be excluded from the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, M.D., PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Depth of Anesthesia
Started | 60
Completed | 59
Not Completed | 1
Not completed — Device did not record data | 1

BASELINE CHARACTERISTICS:
Arm/Group | Depth of Anesthesia
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  Black or African American | 7
  White | 43
  Hispanic or Latino | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Movements as Response to Laryngeal Mask Airway (LMA) Insertion
Description: Correlation between qNOX-qNOX and rough clinical signs of insufficient anti-nociception during Laryngeal Mask Airway (LMA) insertion The Laryngeal Mask Airway (LMA) insertion occurs during the induction, lasting an average of 5-10 minutes.
  Total number of movements reported for the group as a whole and not per participant.
Time Frame: Approximately 10 minutes
Measure: Number; unit: Number of Movements for the whole group
Arm/Group | Depth of Anesthesia
Number analyzed (Participants) | 59
Number of Movements for the whole group | 16

2. Primary Outcome: Number Coughing/Bucking
Description: Coughing/bucking as a response to intraoperative stimuli. The total number of coughing/bucking reported intraoperatively for the group as a whole was recorded.
  The intraoperative period lasted approximately 30 min to 3 hours.
Time Frame: Intraoperative period (30 minutes to 3 hours)
Measure: Number; unit: Number of intraop coughing/bucking
Arm/Group | Depth of Anesthesia
Number analyzed (Participants) | 59
Number of intraop coughing/bucking | 21

3. Secondary Outcome: Number of Intraoperative Movements
Description: Movements as a response to intraoperative stimuli. The total number of movements reported intraoperatively for the group as a whole was recorded.
  The intraoperative period lasted approximately 30 min to 3 hours.
Time Frame: Intraoperative period (30 minutes to 3 hours)
Measure: Number; unit: number of intraop movements
Groups:
- Depth of Anesthesia: Each subject will have the qCON-qNOX monitor on his/her forehead + the BIS monitor
Arm/Group | Depth of Anesthesia
Number analyzed (Participants) | 59
number of intraop movements | 21

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Depth of Anesthesia: Each subject will have the BIS monitor on his/her forehead + the qCON-qNOX monitor
Arm/Group | Depth of Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT02928172/Prot_SAP_000.pdf